CLINICAL TRIAL: NCT06670469
Title: The Effect of Flipped Learning and Escape Room Method on Nursing Students' Infection Control Knowledge and Learning Skills: a Randomized Controlled Study
Brief Title: Flipped Learning and Escape Room Method on Nursing Students
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Aysun Acun 9
Record Dates: First submitted 2024-10-24; First posted 2024-11-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Nursing Students
Keywords: Escape room; Flipped learning; Infection control; Nursing Students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- nursing students: Education of nursing students

SUMMARY:
The impact of interactive education methods on nursing education will be evaluated.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of reverse learning and escape room methods on nursing students' infection control knowledge and learning skills. The study is an original study in terms of focusing on infection control with relevant interactive methods. The study will contribute to the literature in terms of the development of knowledge-based skills such as providing hand hygiene, opening sterile bundles, opening and placing sterile materials in sterile bundles, wearing and removing personal protective equipment, and disposing of waste materials within the scope of infection control. In addition, the questions to be answered in the study are listed below.

ELIGIBILITY:
Inclusion Criteria:

* Receiving training on infection control for the first time

Exclusion Criteria:

* Having received training on infection control before
* Not attending the final test, follow-up test
* Not attending class

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nursing students
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants to measure the rate of influence on knowledge level with reverse learning and escape room teaching methods | 01/11/2024-15/12/2024
  Education level of nursing students

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Seyh Edebali University, Bilecik, Turkey (Türkiye)

REFERENCES:
- [Derived] Acun A, Yildirim A. Learning With Fun: The Effect of Flipped Learning and Escape Room Method on Nursing Students' Infection Control Knowledge and Learning Skills. Int J Nurs Pract. 2025 Oct;31(5):e70067. doi: 10.1111/ijn.70067. PMID 41032006